CLINICAL TRIAL: NCT04045288
Title: SWITCH Implementation Effectiveness Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Collaborators: Kansas State University (Other); University of Nebraska (Other); Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Gregory Welk, Barbara E. Forker Professor of Kinesiology, Iowa State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-68001-23242
Record Dates: First submitted 2019-07-31; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Sedentary Behavior; Health Promotion; Overweight and Obesity; Healthy Lifestyle; Diet, Healthy
Keywords: School Wellness Policy; Professional Development; Comprehensive School Physical Activity Programs; Whole-of-School Intervention; Screen Time; Physical Activity
MeSH Terms: conditions — Sedentary Behavior; Overweight; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Pragmatic Cluster Randomized Controlled Superiority Trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Implementation (Active Comparator): All schools in SWITCH receive training through webinars and an in-person conference to learn about the defining elements and school wellness programming in general. Consistent with the standard implementation, schools were added to the online content management system (CMS) and were given access to an online community of practice (CoP) to interact with other schools / teachers in the study. Schools were provided with resources and program materials (i.e. educational modules, trinkets, posters, etc.) but were given autonomy with regard to how they were used within their school. Weekly updates through the online CMS, the CoP, and via direct email correspondence provided information about the weekly corresponding weekly themes, implementation tips, recommended module activities to incorporate, upcoming evaluation needs, important SWITCH dates, and other program reminders.
  Interventions: Behavioral: Standard Implementation
- Enhanced Implementation (Experimental): The 'Enhanced' implementation strategy provided schools with the same training, access and resources as the standard SWITCH implementation along with more personalized, web-based training based on motivational interviewing (MI) techniques and feedback throughout the implementation process. The supplemental support was provided through participation in two online 'checkpoint sessions' that helped schools self-assess their use of the recommended quality elements and setting-specific best practices. The sessions used principles of motivational interviewing (MI) to promote autonomy and motivation for school change through the process. Schools were also provided with information about how to capitalize on support from local 4H program leaders in their county.
  Interventions: Behavioral: Standard Implementation; Behavioral: Enhanced Implementation

INTERVENTIONS:
Behavioral: Standard Implementation — Schools in the Standard implementation model received web-based training, access to on online education / tracking system and programming resources (modules, posters, trinkets) to facilitate wellness programming in their school. They completed audit tools at the beginning to facilitate goal setting and received weekly emails during the 12-week implementation process.
Behavioral: Enhanced Implementation — Schools in the Enhanced implementation model received the same training, web-access, and programming resources as those in the Standard implementation, but also received enhanced monthly support during implementation from the project team. The supplemental web calls (completed jointly by Extension leaders and SWITCH staff) utilized motivational interviewing to help schools build capacity and to enhance motivation for wellness programming.
  Arms: Enhanced Implementation

SUMMARY:
The SWITCH (School Wellness Integration Targeting Child Health) project is a multi-component intervention designed to support school wellness programming and contribute to youth obesity prevention. Consistent with social-ecological models, SWITCH is designed to reach multiple settings within schools while also facilitating engagement with families and community partners. The program focuses on three distinct behaviors known to impact obesity (i.e., physical activity (PA), sedentary behavior (SB) and fruit and vegetable consumption (FV)) in a creative way by challenging children to "switch what they do, view and chew".

DETAILED DESCRIPTION:
Schools provide an ideal setting for coordinated youth obesity prevention but it has proven difficult to widely disseminate evidence-based programs in a cost-effective way. Multi-component programs that target multiple behaviors and reach multiple settings have been widely recommended in both scientific literature and in public health guidelines documents, but there are few examples of integrated social-ecological approaches that offer promise for broad dissemination.

SWITCH initially began as a controlled childhood obesity intervention trial. A limitation of the original SWITCH program is that the print-based materials made it cost-prohibitive to promote broader dissemination, or to engage other schools. Therefore, the focus of subsequent work focused on developing and testing implementation strategies that would enable SWITCH to be more widely disseminated. In a controlled effectiveness study, we demonstrated that a web-based version had similar utility and outcomes as the print-based program, but effects were directly related to the degree of engagement within the school. Through a USDA-funded project, we developed a novel training method designed to facilitate greater adoption and more effective implementation of SWITCH in schools. The focus in this revised SWITCH model was on helping schools to independently manage the implementation of the evidence-based SWITCH program as part of overall school wellness programming. Thus, we have gradually evolved SWITCH from a school-based intervention conducted through schools to a school wellness training method provided for schools. Schools received

Before moving to broader dissemination efforts it was important to determine the dose of training and support needed to assist schools with implementation. Therefore, the focus of this study was on comparing two different implementation approaches. An enhanced capacity building model that included personalized webinars with school leaders (Enhanced) was compared to a streamlined model based on email communication (Standard). Thus, a key goal is to determine the additive benefit of the enhanced school support relative to the standard implementation. Past work has demonstrated that there is considerable variability in the capacity of schools to take on and lead school wellness programming. Therefore, the analyses also directly examined the moderating influence of school capacity on implementation as well as the impact of implementation on outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All students in schools who completed agreement forms and who formed a three-person core team that attended the conference

Exclusion Criteria:

* All students in schools that did not complete agreement forms, attend the school wellness conference, or form a core team

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1984 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Moderate to Vigorous Physical Activity (minutes / day); Youth Activity Profile (YAP) assessment | Change from baseline to 12 weeks
  The estimate of daily MVPA is obtained from the calibrated , online self-report tool (Youth Activity Profile) built into the web-based content management system. Students complete 5 items capturing school activity and 5 items capturing home activity. The data are then processed using validated algorithms to create estimates of time spent in physical activity behavior.
Sedentary Behavior (hours / day); Youth Activity Profile (YAP) assessment | Change from baseline to 12 weeks
  The estimate of time spent in sedentary behavior (outside of school) is obtained from a calibrated, online self-report tool (Youth Activity Profile) built into the web-based content management system. Students complete 5 items capturing general amounts of sedentary behavior. The data are then processed using validated algorithms to create estimates of time spent in sedentary behavior.
School Capacity for Wellness Programming; School Wellness Readiness Assessment | Change from baseline to 12 weeks
  The assessment of school capacity for wellness programming is obtained at both pre and post time points using the School Wellness Readiness Assessment (SWRA) based on work by Holt et al. (2009). The instrument developed specifically for SWITCH captures Structural barriers (Individual and Organizational) and organizational barriers (Individual and Organizational). The instrument will be completed by the school core teams and the subscale scores will be averaged to create an overall indicator of School Capacity.

SECONDARY OUTCOMES:
Average Weekly Tracking Rate (%); Web-based SWITCH tracking tool | Change from baseline to 12 weeks
  Indicators of school, class and student implementation are obtained by computing engagement and utilization of the web-based SWITCH tracking system. Self-monitoring is a key mediating variable in the SWITCH program, so emphasis in training was placed on helping to promote utilization of the SWITCH tracking system to promote behavior change in the three target behaviors: PA ("do"), SB ("view"), and FV consumption ("chew").
Adherence to Quality Element (average score); Checkpoint Implementation Survey | Change from baseline to 12 weeks
  The Checkpoint Implementation Surveys (CIS) were used in a formative way to guide to evaluate the degree to which schools followed the SWITCH 'quality elements' for overall school implementation. School teams self-reported the degree to which they followed each of the five quality elements using a 3-point scale (none = 1, somewhat = 2, and fully = 3). The average score was used as the overall indicator
Adherence to Best Practices (average score); Checkpoint Implementation Survey | Change from baseline to 12 weeks
  The Checkpoint Implementation Surveys (CIS) were used in a formative way to guide to evaluate the degree to which schools followed the SWITCH 'best practices' in the three targeted settings (classrooms, physical education, and lunchroom). School teams self-reported the degree to which their school followed the 3 best practices in each setting using a 3-point scale (none = 1, somewhat = 2, and fully = 3). The average score is used as an overall indicator.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Welk, PhD, Principal Investigator — Iowa State University
Locations (1):
- Iowa State University, Ames, Iowa, United States

IPD SHARING:
Plan to Share IPD: No